CLINICAL TRIAL: NCT05936086
Title: A Randomized Controlled Study of High-dose Cyclophosphamide Induction Therapy in Adult Patients With HLH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: shifeng Lou (Other)
Responsible Party: Sponsor-Investigator, shifeng Lou, Director, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYNK 04
Record Dates: First submitted 2023-05-30; First posted 2023-07-07 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Hemophagocytic Syndrome
Keywords: Hemophagocytic syndrome（HLH）
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Cyclophosphamide; Etoposide; Dexamethasone; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTX(Cytoxan) group (Experimental)
  Interventions: Drug: Cytoxan; Drug: Dexamethasone
- Normal treatment group (Active Comparator)
  Interventions: Drug: Etoposide; Drug: Dexamethasone; Drug: Cyclosporine (CSA)

INTERVENTIONS:
Drug: Cytoxan — Cytoxan 40mg/kg iv qd x 2days (day 1 and 2);
  Arms: CTX(Cytoxan) group
Drug: Etoposide — etoposide(VP16):150 mg/m2, twice a week, 1-2 weeks; 150mg/m2, once a week for the 3rd to 6th week.
  Other Names: VP16
  Arms: Normal treatment group
Drug: Dexamethasone — Dexamethasone: 10 mg/m2/day, week 1 to 2; 5 mg/m2/d for the 3rd to 4th week; 2.5 mg/m2/ day at week 5-6.
Drug: Cyclosporine (CSA) — Cyclosporine (CSA) 100mg Bid, week 1 to 6 (dosed according to 2004 version).
  Arms: Normal treatment group

SUMMARY:
Adult secondary HLH involves tumors, autoimmune diseases and other causes in addition to infection,Infectious factors, theoretically need different treatment methods for different etiology. But adult HLH itself disease .The situation progresses ferociously, which can cause organ damage and blood coagulation disorder and endanger life quickly, with early mortality (30days).It can be more than 50%. On the other hand, although diagnostic techniques have improved significantly, identifying the cause is still costly Time, such as 1-2 weeks for the pathological diagnosis of lymphoma, leads to more patients losing further treatment due to early death.

The opportunity to heal. Therefore, it is important to explore effective induction therapy for adult HLH. In the majority ,Early (30-day) mortality was as high as 40% after cardiac induction using HLH2004 or CHOP(cyclophosphamide, hydroxydaunomycin, Oncovin, and prednisone) induction. HLH, on the other hand, usually requires prompt treatment before the cause is established. Due to a specific infection HLH can benefit from anti-infective therapy. Therefore, it is necessary to explore more effective induction therapy for adult non-infective HLH.It has very important clinical significance. Adult secondary HLH has the common features of a large number of T cell proliferation and activation and a significant reduction of NK(natural killer) cells, in which the central liNK(natural killer) is a large number of T cells proliferation and secomplete remission etion of cytokines, which can be used as induction therapy.Common target is also the pathological basis for designing unified induction scheme. Cyclophosphamide is a commonly used alkylated chemotherapy drug,It's also an important immunosuppressant. Based on the treatment of regenerative disorders anemia, allogeneic hematopoietic stem cell transplantation prevention.Experience with Plant versus Host disease (GVHD) has shown that the use of cyclophosphamide exceeds a total dose of 25mg/day,Two days can effectively kill CD8(cluster of differentiation 8 )+ or CD4(cluster of differentiation 4

)+T cells, and the maximum tolerated dose of this drug in humans exceeds 50mg/kg/day for two days. Aiming at the central liNK(natural killer) of adult HLH pathogenesis, The investigators designed for the first time to use a large dose of cyclophosphamide (25mg-50mg/kg/day 2days) to inhibit the activation of T cells, inhibit the production of cytokines and block the development mechanism of HLH. This study intends to conduct a randomized controlled study, with HLH2004 scheme as the control, and the observation is large efficacy and safety of dose cyclophosphamide in induction therapy of non-infective adult HLH in order to complete remission eate a new induction Treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 65 years old (including the critical value), gender is not limited;
2. According to the diagnostic criteria of HLH-2004, HLH can be diagnosed if any of the following two criteria are met:

<!-- -->

1. Molecular diagnosis is consistent with HLH: Currently known HLH related pathogenic genes exist, such as PRF1, UNC13D, STX11, STXBP2, Rab27a, LYST, SH2D1A, BIRC4, ITK, AP3β1, MAGT1, CD27 (cluster of differentiation antigen 27 )and other pathological mutations.
2. Meet 5 or more of the following 8 indicators:

   * Fever: body temperature > 38.5 ℃, continuous > 7 d; ② Splenomegaly;

     * Hemocytopenia (involving two or three peripheral blood lines) : hemoglobin < 90 g/L (< 4 weeks infant, hemoglobin < 100 g/L), platelet < 100×109/L, neutrophils < 1.0×109/L and not caused by reduced hematopoietic function of bone marrow; ④ High triglyceride (TG) sepsis and/or low fibrinogenemia: triglyceride > 3 mmol/L or 3 standard deviations above the same age, fibrinogen < 1.5g /L or less than 3 standard deviations for the same age; (5) Hematophagy was found in bone marrow, spleen, liver or lymph nodes;

       * The activity of NK cells is decreased or absent;

         ⑦ Serum ferritin increase: ferritin ≥500 μg/L; Elevated sCD25 (soluble interleukin-2 receptor). (3) Those who can understand the research content, agree to comply with the research plan, and voluntarily sign the informed consent.

Exclusion Criteria:

1. HLH caused by treatable infectious causes (such as bacteria, fungi, viruses (except Epstein-Barr virus), protozoa, etc.);
2. Have a history of allergy or contraindications to the drugs involved in the program;
3. Organ damage caused by long-term chronic diseases;
4. Extreme physical weakness, unstable vital signs and inability to tolerate large doses of cyclophosphamide;
5. Severe and/or uncontrolled co-morbidivities (e.g., uncontrolled diabetes, pulmonary hypertension, etc.) that the investigator believes may pose an unacceptable safety risk or interfere with protocol compliance;
6. Mental instability or history of severe mental illness
7. Other factors determined by the researcher that subjects are not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
complete response rate | up to 30days
  Efficacy evaluation measures included serum sCD25, ferritin, blood count, triglyceride, blood-phagocytosis, and consciousness level (CNS HLH) returning to normal range
Near complete response rate | up to 30days
  Blood routine red blood cells, white blood cells, platelets returned to normal + other laboratory indicators improved by 50%

SECONDARY OUTCOMES:
partial complete response rate | up to 30days
  The antipyretic time, liver function, cytokine concentration, blood image recovery time and other indicators were better than the control group
Single improvement degree among 8 indicators of diagnostic criteria | up to 30days
  Single improvement degree among 8 indicators of diagnostic criteria
30-day mortality rate | up to 30days
  30-day mortality rate
Antipyretic time | up to 30days
  Body temperature is back in the normal range
Invalid (NR) : Complete response and near Complete response are not satisfied, or one of the following conditions occurs | up to 30days
  1. The body temperature did not decrease for three consecutive days, and secondary bacterial or fungal infection could be excluded.
  2. Or continuous deterioration of liver function;
  3. Interleukin-2R and ferritin levels increased continuously.
  4. Coagulation dysfunction continues to worsen.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wen, doctor, Study Director — Hematology Medical Center, the Second Affiliated Hospital of PLA Army Medical University; Huaer Shu, bachelor, Study Director — Chongqing Kaizhou District People's Hospital; Hongbin Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University; Jinglong Lv, master, Study Director — Three Gorges Central Hospital Affiliated to Chongqing University; Zhangqin luo, bachelor, Study Director — Yongchuan Hospital affiliated to Chongqing Medical University; Liang Fang, master, Study Director — Chongqing Ninth People's Hospital; Yizhi Xu, doctor, Study Director — People's Hospital of Chongqing; Zailiang Yang, doctor, Study Director — Fuling Hospital affiliated to Chongqing University
Locations (1):
- The Second affiliated Hosptial of Chongqing medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided